CLINICAL TRIAL: NCT00325871
Title: The Effect of Concurrent Chemoradiation on Circulating Endothelial Progenitor Cells in Colorectal Cancer
Brief Title: Chemoradiation and Endothelial Progenitor Cells in Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yu-Jen Chen, Head, Department of Radiation Oncology, Mackay Memorial Hospital
Other Study IDs: MMH-I-S-243
Record Dates: First submitted 2006-05-12; First posted 2006-05-15 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Procedure: concurrent chemoradiation

SUMMARY:
Colorectal cancer (CRC) is one of the common malignancies worldwide, accounting for a significant percentage of cancer mortality. Concurrent chemoradiation (CCRT) is now a standard treatment for unresectable malignancies of anorectum. To improve quality of life, CCRT is also commonly applied in treatment of lower rectal and anal canal cancer to preserve anal sphincter function. The most commonly used chemotherapeutic drugs combined with radiation as radiosensitizers is 5-fluorouracil (5-FU). Circulating endothelial progenitor cells (EPC), which contribute to the tumor vessel formation, reflect the response to chemotherapy both in animal model and clinical trial. Thus, circulating EPC can be used as a marker for optimizing and monitoring the anti-angiogenesis therapy including angiogenesis inhibitors and chemotherapy. Whether circulating EPC can be served as a marker of CCRT efficacy or not remains undetermined. Since CCRT is now a standard treatment of locally advanced and high-risk CRC, the development of a surrogate marker for monitoring CCRT response and optimize treatment intensity is very important.

In this grant we intent to monitor the levels of circulating EPC in locally advanced and high-risk CRC patients before, during and after CCRT. To further characterize the changes in function and biology of EPC caused by CCRT, a syngeneic animal model will be also used to evaluate the clonogenecity and specific gene expression of EPC in tumor-bearing mice receiving CCRT.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is one of the common malignancies worldwide, accounting for a significant percentage of cancer mortality. The incidence in both developing and developed countries has been increasing over the past few decades (1). Radiation therapy, either as post-operative adjuvant treatment for resectable disease or definitive treatment along with chemotherapy for unresectable disease, has an important role in management of this cancer (1-4).

Concurrent chemoradiation (CCRT) is now a standard treatment for cervical cancer (bulky and locally advanced lesions) (5) and unresectable malignancies of gastrointestinal system origin (esophagus, stomach, pancreas and anorectum) (6-9). To improve quality of life, CCRT is also commonly applied in treatment of lower rectal and anal canal cancer to preserve anal sphincter function (9). The most commonly used chemotherapeutic drugs combined with radiation as radiosensitizers are cis-platinum, 5-fluorouracil (5-FU) and mitomycin C (6-9). These drugs are myelosuppressive and prone to cause life-threatening neutropenia, anemia or thrombocytopenia, which are more severe than those with radiotherapy alone (5-9). To avoid unnecessary over-treatment in CRC, the optimization of CCRT is of critical importance. Herein, the development of a surrogate marker for monitoring treatment efficacy is pivotal to optimize CCRT.

Angiogenesis is a heavily regulated process, which is involved by complex interactions between inhibitory and stimulatory angiogenic factors. It is essential for tumor growth, progression and metastasis and is correlated with poor prognosis in cancer patients including CRC. Many novel compounds that potently inhibit formation of neoplastic blood vessels have been recently developed. There is increasing interest in developing angiogeneis-suppressive agents for colorectal cancer treatment and growing number of anti-angiogenesis drugs currently being evaluated in clinical trials for CRC. Promising results have been reported include an increase in overall survival and reduction in the risk of death (Bevacizumab), reversal of cellular resistance (Cetuximab) and activity as second-line therapy in patients who have exhausted other available treatment options (Cetuximab, ABX-EGF, PTK-787, Gefitinib, Erlotinib) (10,11).

Although the therapeutic role of angiogenesis target therapy has been approved in cancer treatment including CRC, the way to optimize the dose of angiogenesis inhibitors remains to be determined because of the lack of reliable surrogate markers of tumor angiogenesis. Shaked et al. reported that the levels of circulating endothelial progenitor cells (EPC), which contribute to the tumor vessel formation, reflect the anti-tumor efficacy of anti-angiogenesis regimens (12). Growing evidence suggests that the levels of circulating EPC reflect the response to chemotherapy both in animal model and clinical trial (13,14). Thus, circulating EPC can be used as a marker for optimizing and monitoring the anti-angiogenesis therapy including angiogenesis inhibitors and chemotherapy.

Whether circulating EPC can be served as a marker of CCRT efficacy or not remains undetermined. Since CCRT is now a standard treatment of locally advanced and high-risk CRC, the development of a surrogate marker for monitoring CCRT response and optimize treatment intensity, again, is very important.

In this grant we intent to monitor the levels of circulating EPC in locally advanced and high-risk CRC patients before, during and after CCRT. To further characterize the changes in function and biology of EPC caused by CCRT, a syngeneic animal model will be also used to evaluate the clonogenecity and specific gene expression of EPC in tumor-bearing mice receiving CCRT.

References

1. Midgley R, Kerr D. Colorectal cancer. Lancet 1999;353:391-399.
2. Fisher B, Wolmark N, Rockette H, et al. Postoperative adjuvant chemotherapy or radiation therapy for rectal cancer: results from NSABP protocol R-01. J Natl Cancer Inst 1988;80:21-29.
3. O'Connell MJ, Martenson JA, Wieand HS, et al. Improving adjuvant therapy for rectal cancer by combining protracted-infusion fluorouracil with radiation therapy after curative surgery. New Engl J Med 1994;331:502-507.
4. Skarlatos J, Kosma L, Koukourakis M, et al. Hypofractionated radiotherapy with concurrent 5-fluorouracil radiosensitisation for recurrent or locally advanced colorectal cancer. A phase II study. Int J Colore Dis 1996;11:206-210.
5. Rose PG, Bundy BN, Watkins EB, et al. Concurrent cisplatin-based radiotherapy and chemotherapy for locally advanced cervical cancer. New Engl J Med 1999;340:1144-1153.
6. Cooper JS, Guo MD, Herskovic A, et al. Chemoradiotherapy of locally advanced esophageal cancer: long-term follow-up of a prospective randomized trial (RTOG 85-01). Radiation Therapy Oncology Group. J Am Med Assoc 1999;281:1623-1627.
7. Henning GT, Schild SE, Stafford SL, et al. Results of irradiation or chemoirradiation for primary unresectable, locally recurrent, or grossly incomplete resection of gastric adenocarcinoma. Int J Radiat Oncol 2000;46:109-118.
8. Mitchell SE, Mendenhall WM, Zlotecki RA, et al. Squamous cell carcinoma of the anal canal. Int J Radiat Oncol 2001;49:1007-1013.
9. Thomas CR, Weiden PL, Traverso LW, et al. Concomitant intraarterial cisplatin, intravenous 5-flourouracil, and split-course radiation therapy for locally advanced unresectable pancreatic adenocarcinoma: a phase II study of the Puget Sound Oncology Consortium (PSOC-703). Am J Clin Oncol 1997;20:161-165.
10. Kelly H. Goldberg RM. Systemic therapy for metastatic colorectal cancer: current options, current evidence. Journal of Clinical Oncology. 23(20):4553-60, 2005
11. Mancuso A. Sternberg CN. Colorectal cancer and antiangiogenic therapy: what can be expected in clinical practice?. Critical Reviews in Oncology-Hematology. 55(1):67-81, 2005 Jul.
12. Schneider M. Tjwa M. Carmeliet P. A surrogate marker to monitor angiogenesis at last. Cancer Cell. 7(1):3-4, 2005.
13. Bertolini F. Paul S. Mancuso P. Monestiroli S. Gobbi A. Shaked Y. Kerbel RS. Maximum tolerable dose and low-dose metronomic chemotherapy have opposite effects on the mobilization and viability of circulating endothelial progenitor cells. Cancer Research. 63(15):4342-6, 2003.
14. Zhang H. Vakil V. Braunstein M. Smith EL. Maroney J. Chen L. Dai K. Berenson JR. Hussain MM. Klueppelberg U. Norin AJ. Akman HO. Ozcelik T. Batuman OA. Circulating endothelial progenitor cells in multiple myeloma: implications and significance. Blood. 105(8):3286-94, 2005

ELIGIBILITY:
Inclusion Criteria:

* Colorectal cancer patients indicated for chemoradiation

Exclusion Criteria:

* With major systemic disease including other cancer, diabetes, cardiovacular disease.
* Received prior chemotherapy or radiotherapy within 1 month
* Receiving immunosuppressants

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Rectal cancer post-op with CCRT
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2006-04; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Jen Chen, MD, PhD, Principal Investigator — Department of Radiation Oncology, Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin CC, Liu CY, Chen MJ, Wang TE, Chu CH, Wang HY, Shih SC, Hsu ML, Hsu TC, Chen YJ. Profiles of circulating endothelial cells and serum cytokines during adjuvant chemoradiation in rectal cancer patients. Clin Transl Oncol. 2013 Oct;15(10):855-60. doi: 10.1007/s12094-013-1004-6. Epub 2013 Feb 12. PMID 23401019